CLINICAL TRIAL: NCT01160614
Title: An Open-label Study to Characterize the Pharmacokinetics and Safety of Oxycodone Hydrochloride q12h Controlled-Release (ORF) Tablets in Pediatric Patients Aged 6 to 16 Years Inclusive, Who Require Opioid Analgesia
Brief Title: Pharmacokinetics and Safety of ORF Tablets in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OTR1020; 2010-020510-29 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Opioid Analgesia
Keywords: Pediatric; Post-operative; Nonsurgical; patients; Opioid
MeSH Terms: interventions — Open Reading Frames; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ORF Tablets (Experimental): ORF Tablets
  Interventions: Drug: Oxycodone hydrochloride controlled-release (ORF) tablets

INTERVENTIONS:
Drug: Oxycodone hydrochloride controlled-release (ORF) tablets — Oxycodone hydrochloride controlled-release (ORF) tablets (10 mg, 15 mg or 20 mg) taken every 12 hours

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) of single-dose ORF tablets in pediatric patients aged 6 to 16 years, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the parent or legal guardian and patient assent, when appropriate.
* Children of either gender, aged 6 to 16 years, inclusive.
* Have or are expected to have moderate to severe pain for an extended period of time requiring inpatient opioid analgesic treatment for at least 12 hours as this is the minimum duration of study period treatment.
* In order to receive the first oral dose, patients must have respiratory stability, including a sustained SpO2 of at least 92% with or without supplemental oxygen during the 15 minute period just prior to dosing.
* Must be inpatient for the treatment period of the study.
* The patient's anticipated opioid analgesic requirement over the first 12 hours that will follow administration of ORF must be equivalent to at least 10 mg of intravenous (IV) morphine.
* Have adequate pain control during the 6 hours prior to study drug administration, based on appropriate clinical assessment.
* Must be sufficiently alert to communicate and complete the faces pain scales-revised (FPS-R) or 100-mm visual analogue scale (VAS).
* Females who are of child bearing potential must be using an adequate and reliable method of contraception (e.g., barrier with additional spermicidal foam or jelly, intra-uterine device, hormonal contraception) or be abstinent.
* If female, must have a negative pregnancy test and be non-lactating.
* Must be able to swallow tablets whole.
* Must have stable vital signs.
* Must have vascular access to facilitate blood draws.
* Must be willing and able to participate in all aspects of this study involving use of oral medications, patient evaluation, and phlebotomy, as evidenced by written informed consent from the parent or legal guardian and written patient assent when required by the local IRB/EC.
* Must be willing to have up to 10 milliliters (mL) of blood collected for blood analysis (7 mL for primary PK and 3 mL for secondary PK analysis); and up to 10 mL of blood for pre-specified safety laboratory tests, without safety concerns.
* Must be treated with an opioid for a minimum of 96 hours prior to first dose of ORF.

Exclusion Criteria:

* Any history of hypersensitivity or medical contraindication for the use of oxycodone (this does not exclude patients with a history of expected opioid-related adverse events (AEs), such as light-headedness, dizziness, sedation, nausea, or vomiting).
* Any current history of medical or surgical conditions that might significantly interfere with the gastrointestinal absorption, distribution, metabolism, or excretion of oxycodone (this includes any history of serious disease+ of the gastrointestinal tract, liver, kidneys, and/or blood-forming organs).
* Received oxycodone in the 24 hours prior to study drug administration. .
* Received epidural (or regional) anesthesia < 12 hours prior to the first oral dose of ORF.
* A current history of malabsorption syndrome.
* A current diagnosis of sleep apnea within the last year.
* Reduced renal function (serum creatinine > 1.8 X the upper limit of normal for age).
* Hepatic impairment as evidenced by serum alanine amino transferase (ALT) or serum aspartate amino transferase (AST) > 5 times the upper limit of normal (ULN) for age.
* Currently taking any medications which are CYP3A4 inhibitors.
* Impaired respiratory reserve including severe acute or chronic lung disease, or patients receiving mechanical respiratory support, including mechanical ventilation, BIPAP, or CPAP 6 hours prior to the first oral dose and during the entire oral treatment period.
* Impaired cardiovascular stability (e.g., the day of surgery for cardiac surgery patients).
* Participated in a clinical drug study within 30 days preceding the initial dose in this study.
* Patients who have had surgery within 96 hours prior to the day of the first dose of study drug.
* Deemed to be unsuitable by the investigator for reason(s) not specifically stated in the exclusion criteria.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (13):
  - Maricopa Medical Center, Phoenix, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - LS Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital Association, Aurora, Colorado
  - Research Facility, Miami, Florida
  - F3900 C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Akron Children's Hospital, Akron, Ohio
  - The Children's Hospital at OUMC, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Med Center of Dallas, Dallas, Texas
  - Scott & White Memorial Hospital & Clinic, Temple, Texas
  - University of Washington School of Medicine - Harborview Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Royal Children's Hospital, Parkville, Australia
- Finland (2):
  - Helsinki University Central Hospital/Children and Adolescent Hospital, Helsinki
  - Kuopio University Hospital/Operative Services and Intensive Care, Kuopio
- Waikato Clinical Research (2008) Ltd, Hamilton, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit: 18-Aug-2010; Last Patient Last Visit: 16-Aug-2011. The study was conducted at 11 sites in the United States and Australia.
Pre-assignment Details: Pediatric patients who were anticipated to have pain requiring opioid analgesia.
Groups:
- 6 to < 12 Years: Children aged 6 to < 12 Years received ORF Tablets (10 mg, 15 mg or 20 mg taken every 12 hours). Study treatment could have lasted from 12 hours (single dose) to 72 hours (5 doses).
- ≥ 12 to ≤ 16 Years: Children aged ≥ 12 to ≤ 16 Years received ORF Tablets (10 mg, 15 mg or 20 mg taken every 12 hours). Study treatment could have lasted from 12 hours (single dose) to 72 hours (5 doses).
Period: Overall Study
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Started | 5 | 25
Completed | 5 | 23
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years | Total
Number analyzed (Participants) | 5 | 25 | 30
Age Continuous [Mean (Standard Deviation); unit: Years] | 10.6 (0.9) | 14.1 (1.6) | 13.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 14 | 17
  Male | 2 | 11 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 4 | 21 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Single-dose PK Metric: Area Under the Plasma Concentration-time Curve From Hour 0 to the Last Measurable Plasma Concentration [AUCt]
Time Frame: Up to 24 hours
Population: The full analysis population for PK (N = 30) was defined as patients who received at least 1 dose of oral study drug and had at least 1 valid quantifiable PK metric
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- 6 to < 12 Years (10 mg ORF): Children from 6 to < 12 years received a single dose of 10 mg ORF
- 6 to < 12 Years (15 mg ORF): Children from 6 to < 12 years received a single dose of 15 mg ORF
- 6 to < 12 Years (20 mg ORF): Children from 6 to < 12 years received a single dose of 20 mg ORF
- ≥ 12 to ≤ 16 Years (10 mg ORF): Children from ≥ 12 to ≤ 16 years received a single dose of 10 mg ORF
- ≥ 12 to ≤ 16 Years (15 mg ORF): Children from ≥ 12 to ≤ 16 years received a single dose of 15 mg ORF
- ≥ 12 to ≤ 16 Years (20 mg ORF): Children from ≥ 12 to ≤ 16 years received a single dose of 20 mg ORF. One patient took a single dose of ORF 30 mg and is included in this dose level.
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 8
ng*h/mL | 129.2 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 121.1 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 272.2 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 85.5 (39.3) | 193.0 (149.4) | 264.4 (128.1)

2. Primary Outcome: Single-dose PK Metric: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (AUCinf)
Description: Due to insufficient sampling, AUCinf was not estimated.
Time Frame: Up to 24 hours
Reporting Status: Not Posted

3. Secondary Outcome: Multiple-dose PK Metric: Minimum Observed Plasma Concentration Just Prior to the Next Dose (Cmin)
Time Frame: Up to 72 hours if all 5 doses were administered
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 6 to < 12 Years (10 mg ORF): Children from 6 to < 12 years who received multiple doses of 10 mg ORF
- 6 to < 12 Years (15 mg ORF): Children from 6 to < 12 years who received multiple doses of 15 mg ORF
- 6 to < 12 Years (20 mg ORF): Children from 6 to < 12 years who received multiple doses of 20 mg ORF
- ≥ 12 to ≤ 16 Years (10 mg ORF): Children from ≥ 12 to ≤ 16 years who received multiple doses of 10 mg ORF
- ≥ 12 to ≤ 16 Years (15 mg ORF): Children from ≥ 12 to ≤ 16 years who received multiple doses of 15 mg ORF
- ≥ 12 to ≤ 16 Years (20 mg ORF): Children from ≥ 12 to ≤ 16 years who received multiple doses of 20 mg ORF. One patient took a single dose of ORF 30 mg and is included in this dose level.
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 1 | 1 | 0 | 3 | 4 | 3
ng/mL | 15.5 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 17.3 (NA) — Standard deviation not calculable since there was only 1 patient in this group |  | 4.8 (1.9) | 11.9 (6.9) | 19.1 (2.7)

4. Primary Outcome: Single-dose PK Metric: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 8
ng/mL | 12.3 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 16.6 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 21.9 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 8.3 (1.9) | 26.6 (16.0) | 26.2 (7.9)

5. Primary Outcome: Single-dose PK Metric: Time to Maximum Plasma Concentration (Tmax)
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 8
hour (h) | 6 [6 to 6] | 3 (NA) [3 to 3] | 12 (NA) [12 to 12] | 5.3 (1.011) [4.6 to 6] | 3 (1.26) [1.5 to 4.5] | 6 (6.663) [4.4 to 24.1]

6. Primary Outcome: Single-dose PK Metric: Apparent Terminal Phase Rate Constant (Lamda z)
Description: Due to insufficient sampling, Lamda z was not estimated.
Time Frame: Up to 24 hours
Reporting Status: Not Posted

7. Primary Outcome: Single-dose PK Metric: Apparent Plasma Terminal Phase Half/Life (t1/2z)
Description: Due to insufficient sampling, t1/2z was not estimated.
Time Frame: Up to 24 hours
Reporting Status: Not Posted

8. Primary Outcome: Single-dose PK Metric: Lag Time Was Estimated as the Time Point Immediately Prior to the First Measurable Plasma Concentration Value (Tlag)
Description: Due to insufficient sampling, tlag was not estimated.
Time Frame: Up to 24 hours
Reporting Status: Not Posted

9. Primary Outcome: Single- and Multiple-dose PK Metric: Mean Area Under the Plasma Concentration During Each Dosing Interval-time Curve From Hour 0 to 12 Hours of the First Dose of ORF (AUC 0-12)
Time Frame: Up to 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- 6 to < 12 Years (10 mg ORF): Children from 6 to < 12 years who received single or multiple doses of 10 mg ORF
- 6 to < 12 Years (15 mg ORF): Children from 6 to < 12 years who received single or multiple doses of 15 mg ORF
- 6 to < 12 Years (20 mg ORF): Children from 6 to < 12 years who received single or multiple doses of 20 mg ORF
- ≥ 12 to ≤ 16 Years (10 mg ORF): Children from ≥ 12 to ≤ 16 years who received single or multiple doses of 10 mg ORF
- ≥ 12 to ≤ 16 Years (15 mg ORF): Children from ≥ 12 to ≤ 16 years who received single or multiple doses of 15 mg ORF
- ≥ 12 to ≤ 16 Years (20 mg ORF): Children from ≥ 12 to ≤ 16 years who received single or multiple doses of 20 mg ORF. One patient took a single dose of ORF 30 mg and is included in this dose level.
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 2 | 2 | 1 | 4 | 8 | 9
ng*h/mL | 67.5 (29.1) | 114.5 (9.4) | 112.8 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 82.5 (13.4) | 139.0 (105.2) | 174.2 (112.7)

10. Primary Outcome: Single- and Multiple-dose PK Metric: Maximum Observed Plasma Concentration From Hour 0 to 12 Hours of the First Dose of ORF (Cmax 0-12)
Time Frame: Up to 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 9 | 11
ng/mL | 9.4 (4.2) | 23.5 (9.8) | 21.9 (NA) — Standard deviation not calculable since there was only 1 patient in this group | 10.0 (2.3) | 21.8 (14.2) | 25.1 (14.2)

11. Primary Outcome: Single- and Multiple-dose PK Metric: Time to Maximum Plasma Concentration From Hour 0 to 12 Hours of the First Dose of ORF (Tmax 0-12)
Time Frame: Up to 12 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 6 to < 12 Years (10 mg ORF) | 6 to < 12 Years (15 mg ORF) | 6 to < 12 Years (20 mg ORF) | ≥ 12 to ≤ 16 Years (10 mg ORF) | ≥ 12 to ≤ 16 Years (15 mg ORF) | ≥ 12 to ≤ 16 Years (20 mg ORF)
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 9 | 11
h | 9 (4.243) [6 to 12] | 7.3 (6.131) [3 to 11.7] | 12 (NA) [12 to 12] | 4.6 (3.526) [2.8 to 12] | 4.5 (3.036) [1.5 to 12] | 6 (2.931) [3.3 to 11.9]

12. Primary Outcome: Single- and Multiple-dose PK Metric: Lag Time Estimated as the Time Point Immediately Prior to the First Measurable Plasma Concentration Value From Hour 0 to 12 Hours of the First Dose of ORF (Tlag 0-12)
Description: Due to insufficient sampling, tlag 0-12 was not estimated.
Time Frame: Up to 12 hours
Reporting Status: Not Posted

13. Primary Outcome: The Number of Patients With Adverse Events as a Measure of Safety
Time Frame: Adverse events (AEs) & serious adverse events (SAEs) were reported from start of study participation through the period beyond study completion (AEs) & through 30 days following last study drug dose, or until last study visit, whichever was later (SAEs).
Population: The safety population (N = 30) was defined as the group of patients who received study drug
Measure: Number; unit: participants
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 5 | 25
participants
  Death | 0 | 0
  Serious Adverse Event (SAE) | 0 | 1
  Any TEAE reported in ≥ 5% of participants | 5 | 16

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) & serious adverse events (SAEs) were reported from start of study participation through the period beyond study completion (AEs) & through 30 days following last study drug dose, or until last study visit, whichever was later (SAEs).
Description: AEs were learned of through spontaneous reports or patient interview.
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/25
Other Adverse Events (participants affected / at risk) | 5/5 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 to < 12 Years (N=5) | ≥ 12 to ≤ 16 Years (N=25)
Medical device complication (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 to < 12 Years (N=5) | ≥ 12 to ≤ 16 Years (N=25)
Constipation (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 5
Oxygen saturation decreased (Investigations) | 0 | 2
Respiratory rate decreased (Investigations) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 1
Sedation (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days